CLINICAL TRIAL: NCT05090228
Title: Right Ventricle REmodeling After Pulmonary vAlve Replacement and Percutaneous Pulmonary Valve InseRtion, a Functional and Histopathological Assessment
Brief Title: Right Ventricle Remodeling After Pulmonary Valve Replacement and Percutaneous Pulmonary Valve Insertion
Acronym: RV-REPAIR
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Michiel Voskuil, MD, PhD, M. Voskuil, MD, PhD, UMC Utrecht
Other Study IDs: NL53771.041.15; 15-448/M (Other: METC UMC_Utrecht)
Record Dates: First submitted 2015-12-03; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Endomyocardial Fibrosis; Pulmonary Valve Stenosis; Pulmonary Valve Insufficiency
Keywords: Right ventricle (reverse) remodeling (fibrosis); Right ventricle pressure overloading; Right ventricle volume overloading
MeSH Terms: conditions — Endomyocardial Fibrosis; Pulmonary Valve Stenosis; Pulmonary Valve Insufficiency; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for biomarker studies. Endomyocardial biopsies for (diffuse) fibrosis studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PVR/PPVI: Adult patients with congenital heart disease (GUCH) undergoing pulmonary valve replacement (PVR) or percutaneous pulmonary valve insertion (PPVI).

SUMMARY:
This study investigates damage of the right cardiac chamber in adult patients with a congenital heart defect involving the pulmonary valve (the heart valve between the right cardiac chamber and the lungs). The investigators want to investigate if novel, less invasive techniques are feasible to assess damage of this right cardiac chamber, to improve follow-up and timing of intervention (valve replacement) in this group of patients.

DETAILED DESCRIPTION:
Rationale:

In congenital heart disease the right heart is often affected, in contrast to acquired heart disease where the left ventricle and left sided valves are most often affected. In congenital patients, the right heart problem is most common linked to dysfunction of the pulmonary valve. In these congenital patients, with defects such as Tetralogy of Fallot (ToF), Double Outlet Right Ventricle (DORV), Pulmonary Valve Atresia, and Ventricular Septum Defect (VSD), the primary origin of the problem are dysplastic Pulmonary Valves (PV) and Right Ventricle Outflow Tract Obstruction (RVOTO). Often these valves or obstructions are excised to be replaced directly or in a later stage. Until the end '90s common therapy was to cut out the pulmonary valve and leave patients without pulmonary valve for 10 to 20 years. This resulted in a pendular flow between right ventricle and pulmonary arteries. This works because the pulmonary vascular resistance is low and therefore inflow is easy. There is also a congenital group in which the primary problem was left sided, but a right-sided problem is created by therapy. Since 20 years the Ross procedure is used for congenital aortic valve stenosis. The pulmonary valve is used in childhood to replace the aortic valve, and needs to be replaced in adolescence by a homograft (graft with human donor valve).

In both these groups (repeat) pulmonary valve replacement is necessary, at some stage, with an open procedure; Pulmonary Valve Replacement (PVR) or catheter procedure; Percutaneous Pulmonary Valve Insertion (PPVI), a method available since 2000. Because these valves only last for 10 to 20 years, timing of intervention is very important.

The last 10 years efforts have been done to delineate the best moment for pulmonary valve replacement. The aim is to prevent right ventricular failure due to pressure overload (stenosis of homograft), volume overload (absence of PV after excision or insufficiency of homograft) or a combination of pressure- and volume-overload, which is believed to be most malignant. In the past emphasis was paid to onset of symptoms instead of preventing right ventricular damage. Because symptoms in right ventricular failure are linked to the 'point of no return' (when the right ventricle doesn't fully recover after pulmonary valve replacement), most likely a better strategy is to intervene before symptoms arise. To be able to make reliable criteria for valve replacement we need to better understand the anatomical and functional impairments of the right ventricle and link this to histopathological changes. The investigators believe myocardial fibrosis is correlated to this 'point of no return'. In the last decades knowledge concerning RV volumes and function, electrocardiographic and exercise capacity has grown. But, the relation between volumes, function and histopathology is missing.

Objective:

Primary objectives: to investigate functional and histopathological changes of the right ventricle before and after PVR or PPVI. To investigate if non-invasive assessment of RV-remodeling including CMR-T1rho mapping is possible and validate this with the golden standard of histopathology.

Secondary objectives: to investigate changes in parameters, using echocardiography, electrocardiography, biomarkers, exercise capacity and quality of life in patients undergoing PVR or PPVI.

ELIGIBILITY:
Inclusion Criteria:

* Individual should meet the European Society of Cardiology criteria for pulmonary valve intervention according to congenital heart disease guidelines.
* Individual has an indication for PVR or PPVI according to the local GUCH heart team
* Individual is ≥18 years of age.
* Individual agrees to have all study procedures performed, and is competent and willing to provide written informed consent to participate in this clinical study.
* Patients are acceptable candidates for PVR or PPVI treatment in accordance with manufacturer's instructions for use.

Exclusion Criteria:

* Individual is younger than 18 years of age.
* Individual has an estimated glomerular filtration rate (eGFR) of <30mL/min/1.73m2, using the MDRD (Modification of Diet in Renal Disease) calculation.
* Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, haemophilia, significant anaemia).
* Individual is pregnant, nursing or planning to be pregnant.
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Individual is currently enrolled in an investigational drug or device trial.
* Individual with any contraindications for MRI:

  1. The presence of implanted non-MRI-compatible cardiac pacemaker or implanted cardioverter defibrillator.
  2. Implanted electronic devices like cochlear implants and nerve stimulators.
  3. Patients who are unable to fit into the bore of the magnet.
  4. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with congenital heart disease with severe Pulmonary Insufficiency and/or Pulmonary Stenosis with an indication for PVR or PPVI.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
histopathology: percentage of fibrosis in biopsies. | 6 months
  endomyocardial biopsies performed during valve replacement RV endomyocardial biopsies performed during valve replacement procedure.
T1 time in ms | before and 6 months after valve replacement
  CMR
T1 rho time in ms | before and 6 months after valve replacement
  CMR
Late gadolinium enhancement | before and 6 months after valve replacement
  CMR

SECONDARY OUTCOMES:
Echocardiographic parameters | before valve replacement and direct post-intervention, 1month and 6 months post-intervention
  Right ventricular strain-rate (1/s).
Electrocardiographic sign of RV hypertrophy | before and 6 months after valve replacement (ECG and Holter)
  Right axis deviation of +110° or more.
Biomarkers | Before and 6 months after valve replacement
  Brain natriuretic peptide (pmol/L)
Quality of life SF-36 | before and 6 months after valve replacement
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Voskuil, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands